CLINICAL TRIAL: NCT04682717
Title: Perfusion Index as a Predictor of Hypotension Following Propofol Induction of General Anesthesia in Geriatric Patients - A Prospective Observational Study.
Brief Title: Perfusion Index as a Predictor of Postinduction Hypotension of General Anesthesia in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Lecturer of anesthesia, Cairo University
Other Study IDs: N-12/2020
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Hypotension on Induction
Keywords: geriatris; postinduction hypotension; perfusion index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- PI group: A cut-off value of baseline PI below which hypotension at 5 min post induction could be predicted will be the primary outcome, while positive and negative predictive values at 15 minutes will be secondary outcomes.
  Interventions: Device: perfusion index monitoring for postinduction hypotension

INTERVENTIONS:
Device: perfusion index monitoring for postinduction hypotension — Hemodynamic parameters will be recorded at 1-min intervals till 10 min after intubation. Hypotension will be defined as a drop in SBP to <30% of baseline or absolute MAP <60 mmHg. MAP <55 mmHg (severe hypotension) will be treated immediately by rapid intravenous fluid administration (10 ml/kg) and ephedrine sulphate 6 mg IV boluses. Bradycardia will be defined as HR <50 bpm or decrease by more than 30% below baseline value, whichever will be lower and will be treated with atropine 0.6 mg IV boluses. The incidence of hypotension will be calculated in 2 sets - 5 min after induction of anesthesia (effect of induction agent) and first 15 min after induction (effect of induction process and endotracheal intubation).

SUMMARY:
The influence of hemodynamic aberrations during anesthesia on adverse outcomes is an important clinical issue. There is evidence that hypotension and hypertension during general anesthesia are independently associated with adverse outcomes in patients having both noncardiac and cardiac surgery.One of the intervals of general anesthesia during which hypotension is prevalent is the period after the induction of anesthesia but before the onset of surgical stimulation. This period is particularly prone to decreased vigilance with regard to hemodynamic changes.

Statistically significant predictors of hypotension 0-10 min after anesthetic induction included: ASA III-V, baseline MAP <70 mm Hg, age > or =50 years, the use of propofol for induction of anesthesia, and increasing induction dosage of fentanyl.While the potential preoperative factors associated with hypotension 5-10 min after the induction of anesthesia in patients with ASA I-II included baseline MAP 70 mm Hg, age > 50 years, use of propofol during induction, and magnitude of fentanyl dose during induction.

Perfusion index (PI) is a relatively new parameter estimating the pulsatility of blood in the extremities, calculated using infrared spectrum as part of plethysmography waveform processing. It is a simple,cost-effective and non-invasive method of assessing peripheral perfusion determined by the percentage of pulsatile to non-pulsatile blood flow in the extremities. PI indicates the status of the microcirculation which is densely innervated by sympathetic nerves, and therefore, is affected by multiple factors responsible for vasoconstriction or vasodilatation of the microvasculature.It is an indicator of systemic vascular resistance (SVR).

PI is said to be useful in monitoring depth of anesthesia, hypothermia, successful epidural placement in parturients, adequate relief from ureteric obstruction, response to fluid therapy in critically ill and intraoperative patients and adequacy of circulation in newborn.The value of PI is inversely related to the vascular tone, though not in a linear fashion. Therefore, vasodilatation reflecting higher baseline PI has been associated with reductions in blood pressure (BP) following spinal anesthesia.The resting SVR can influence incidence and severity of post-spinal hypotension in parturients.

It has been established that a positive correlation between pre-anesthetic plethysmographic variability index (PVI) and reduction in BP following induction of anesthesia using propofol in healthy adults, that is, higher PVI was associated with more mean arterial pressure (MAP) reductions. Similarly, a significant proportion of hypotension after induction of anesthesia with propofol can be attributed to the baseline SVR.

Mehandale SG. and Rajasekhar P. underwent A prospective observational study on fifty adults for the use of Perfusion index as a predictor of hypotension following propofol induction and revealed that a baseline PI <1.05 predicted incidence of hypotension at 5 min with sensitivity 93%, specificity 71%, positive predictive value (PPV) 68% and negative predictive value (NPV) 98%.

the hypothesised was that it is possible to define a threshold baseline value of PI that predicts hypotension based on individual's pre-induction SVR in patients > 65 years old following anesthetic induction with propofol and fentanyl as multifactorial risk for postinduction hypotension.

Outcomes:

A cut-off value of baseline PI below which hypotension at 5 min post induction could be predicted will be the primary outcome, while positive and negative predictive values at 15 minutes will be secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged > 65 years
* belonging to the American Society of Anesthesiologists' Physical Status I to II
* elective surgery under general anesthesia

Exclusion Criteria:

* hypertension,
* vasoactive medications,
* difficult airway

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Thirty patients aged > 65 years undergoing elective surgery under general anesthesia performed in general surgery theater at Kasr Al-Ainy hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
perfusion index | 5 minutes postinduction
  A cut-off value of baseline PI below which hypotension post induction could be predicted

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospitals, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] Jain U, Laflamme CJ, Aggarwal A, Ramsay JG, Comunale ME, Ghoshal S, Ngo L, Ziola K, Hollenberg M, Mangano DT. Electrocardiographic and hemodynamic changes and their association with myocardial infarction during coronary artery bypass surgery. A multicenter study. Multicenter Study of Perioperative Ischemia (McSPI) Research Group. Anesthesiology. 1997 Mar;86(3):576-91. doi: 10.1097/00000542-199703000-00009. PMID 9066323
- [Background] Loeb RG. A measure of intraoperative attention to monitor displays. Anesth Analg. 1993 Feb;76(2):337-41. PMID 8424512
- [Background] Reich DL, Hossain S, Krol M, Baez B, Patel P, Bernstein A, Bodian CA. Predictors of hypotension after induction of general anesthesia. Anesth Analg. 2005 Sep;101(3):622-628. doi: 10.1213/01.ANE.0000175214.38450.91. PMID 16115962
- [Background] van Genderen ME, Bartels SA, Lima A, Bezemer R, Ince C, Bakker J, van Bommel J. Peripheral perfusion index as an early predictor for central hypovolemia in awake healthy volunteers. Anesth Analg. 2013 Feb;116(2):351-6. doi: 10.1213/ANE.0b013e318274e151. Epub 2013 Jan 9. PMID 23302972